CLINICAL TRIAL: NCT07079891
Title: Association Between Ambient Temperature and Myocardial Injury After Noncardiac Surgery in Adults: a Retrospective Single-center Cohort Study
Brief Title: Association Between Ambient Temperature and Myocardial Injury After Noncardiac Surgery in Adults
Status: Completed | Type: Observational
Sponsor: Hao Li (Other)
Responsible Party: Sponsor-Investigator, Hao Li, Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: 20256030
Record Dates: First submitted 2025-06-30; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: MINS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- moderate heat (22.8℃-29.2℃)
  Interventions: Other: MINS
- extreme heat (≥29.2℃)
  Interventions: Other: MINS
- extreme cold (≤-3.5℃)
  Interventions: Other: MINS
- moderate cold (-3.5℃-22.8℃)
  Interventions: Other: MINS

INTERVENTIONS:
Other: MINS — MINS

SUMMARY:
This single-center retrospective cohort study enrolled patients aged ≥18 years who underwent noncardiac surgery between January 2014 and December 2023. The exposure variable was the 7-day average preoperative ambient temperature in Beijing. Univariate and multivariate logistic regression models were used to evaluate the association between temperature and MINS. Inverse probability of treatment weighting (IPTW) analysis was performed to enhance the robustness of the findings. Subgroup analyses were performed across predefined clinical strata.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* underwent noncardiac surgery under general anesthesia

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) classification V;
* outpatient, hysteroscopic, or body surface surgeries
* surgery duration ≤30 min
* absence of postoperative high-sensitivity troponin T (hs-TnT) testing within 30 days
* incomplete clinical data (≥20% missing data)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This retrospective single-center cohort study included 143,095 adult (≥18 years) patients who underwent noncardiac surgery under general anesthesia between January 2014 and December 2023. The exclusion criteria were as follows: (1) American Society of Anesthesiologists (ASA) classification V; (2) outpatient, hysteroscopic, or body surface surgeries; (3) surgery duration ≤30 min; (4) absence of postoperative high-sensitivity troponin T (hs-TnT) testing within 30 days; and (5) incomplete clinical data (≥20% missing data).
Sampling Method: Non-Probability Sample
Enrollment: 143095 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of MINS | POSTOPERATIVE 30 DAYS